CLINICAL TRIAL: NCT03101501
Title: A Prospective Study To Evaluate The Raindrop Near Vision Inlay In Presybopic or Pseudophakic Patients Treated With Mitomycin C Following Femtosecond Flap Creation.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The manufacturing company of the Raindrop Corneal Inlay has stopped distribution or sales of the product.
Sponsor: Key-Whitman Eye Center (Other)
Responsible Party: Principal Investigator, Jeffrey Whitman, MD, President and Chief Surgeon, Key-Whitman Eye Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P17-001
Record Dates: First submitted 2017-03-30; First posted 2017-04-05 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MMC for fibrosis prevention (Experimental): no intervention is required after procedure is performed
  Interventions: Drug: Mitomycin c; Device: Raindrop Near Vision Inlay

INTERVENTIONS:
Drug: Mitomycin c — Low dose mitomycin C at a concentration of 0.02% will be applied a duration of 10 to 30 seconds at the time of the surgical procedure.
Device: Raindrop Near Vision Inlay — Implanted to improve near vision in Presbyopic or Pseudophakic subjects.

SUMMARY:
The clinical objective of this study is to evaluate the Raindrop® Near Vision Inlay for the improvement of near vision in presbyopic or pseudophakic patients treated with low dose Mitomycin C immediately following femtosecond flap creation.

DETAILED DESCRIPTION:
The scientific objective of this study is to evaluate the postoperative incidence of corneal reaction in patients treated with low dose Mitomycin C, immediately following femtosecond flap creation (LASIK correction if needed), and before implantation with the Raindrop corneal inlay in the non-dominant eye. The postoperative incidence of haze, visible by broad tangential illumination of the slit lamp, is known to adversely impact the safety and efficacy of the Raindrop corneal inlay. Three main strategies have been employed to minimize haze incidence after surgery: (i) perfection of the surgical technique, (ii) deeper implantation in the cornea, and (iii) extension of the steroid regimen after surgery. Haze has also been observed after another type of corneal refractive procedure, Photorefractive Keratectomy (PRK). Several prospective studies have shown that Mitomycin C, applied immediately following the PRK laser procedure, is effective in reducing the postoperative incidence of haze.

ELIGIBILITY:
Inclusion Criteria:

4.2.1 Presbyopic patients 41-65 years of age.

4.2.2 Pseudophakic patients at least 50 years of age.

4.2.3 Patients require a near reading add from +1.50 to +2.50 D in the non-dominant eye.

4.2.4 Patients have a photopic pupil size of at least 3.0 mm in the non-dominant eye.

4.2.5 Patients have a corneal thickness greater than or equal to 500 microns in the non-dominant eye.

4.2.6 Patients have corrected distance and near visual acuity of 20/25 or better in each eye.

4.2.7 Patients have distance corrected near visual acuity of 20/40 or worse in each eye.

4.2.8 Patients have no more than a 0.75 D difference at preop between MRSE and cycloplegic refraction spherical equivalent determined at the spectacle plane of each eye.

4.2.9 Patients have targeted MRSE from -0.5 to +1.0 D in the non-dominant eye, with no more than 0.75 D of manifest cylinder with or without LASIK.

4.2.10 Patients are willing and able to sign a written Informed Consent Form prior to any study-specific procedures.

4.2.11 Pseudophakic patients must be at least 3 months after cataract surgery.

4.2.12 Pseudophakic patients must have clear posterior capsule, open posterior capsule (post YAG Capsulotomy), or posterior capsule opacification that is not clinically significant at the opinion of the investigator.

4.2.13 Patients are willing and able to return for scheduled follow-up examinations for 24 months after the corneal inlay surgery.

Exclusion Criteria

4.3.1 Patients with prior corneal surgery including LASIK surgery in the non-dominant eye. (Not including Astigmatic Keratotomy or Limbal Relaxing Incisions)

4.3.2 Patients with clinically significant dry eye (i.e., significant diffuse punctate staining with fluorescein and a tear breakup time less than 8 s) in either eye.

4.3.3 Patients with a planned corneal residual bed thickness that is less than 300 microns (corneal thickness - (intended ablation depth + intended flap thickness)).

4.3.4 Patients with clinically significant macular pathology based on dilated fundus exam and/or optical coherence tomography (OCT) image.

4.3.5 Patients who would be co-managed by an ophthalmologist or optometrist who is not an approved sub-investigator.

4.3.6 Patients with ocular pathology or disease (including pupil pathology such as fixated pupils) that might confound the outcome or increase the risk of adverse event in the investigator's opinion.

4.3.7 Patients taking systemic or topical medications that might confound the outcome or increase the risk of adverse event. Patients taking isotretinoin or amiodarone hydrochloride and any other medication that affects the tear film or accommodation, including but not limited to, mydriatic, cycloplegic and mitotic agents, or any other medications in the investigator's opinion.

4.3.8 Patients with known sensitivity to any planned study medications.

4.3.9 Patients with residual, recurrent, active or uncontrolled eyelid disease.

4.3.10 Patients with significant corneal asymmetry or irregular topography.

4.3.11 Patients with clinically significant anterior segment pathology.

4.3.12 Patients with any corneal abnormality, including but not limited to, slit lamp findings for corneal staining Grade 3 or higher, recurrent corneal erosion or severe basement membrane disease, and pterygium extending onto the cornea.

4.3.13 Patients with ophthalmoscopic/topographic signs of keratoconus or those who are keratoconus suspect.

4.3.14 Patients with history of Herpes zoster or Herpes simplex keratitis.

4.3.15 Pseudophakic patients that have anterior chamber IOLs, multifocal IOLs, or extended range of vision IOLs in either eye.

4.3.16 Patients with any progressive retinal disease or subjects with a history or evidence of retinal vascular occlusion and/or hypercoagulability, because of the risks associated with high pressures during suction application.

4.3.17 Patients with known history of steroid-responsive intraocular pressure increases, glaucoma, preoperative IOP > 21 mm Hg, or are otherwise suspected of having glaucoma.

4.3.18 Patients with amblyopia or strabismus or those who are at risk for developing strabismus postoperatively as determined by corneal light reflex and cover-uncover testing.

4.3.19 Patients with diabetic retinopathy, collagen, vascular, diagnosed autoimmune disease (e.g., lupus, rheumatoid arthritis, fibromylagia), immunodeficiency (e.g., HIV), connective tissue disease, or clinically significant atopic syndrome.

4.3.20 Patients on chronic systemic corticosteroid or other immunosuppressive therapy that may affect wound healing at the opinion of the investigator.

4.3.21 Patients with any type of active cancer (ophthalmic or non-ophthalmic).

4.3.22 Patients with uncontrolled infections of any kind.

4.3.23 Patients who are pregnant, lactating, of child-bearing potential and not practicing a medically approved method of birth control, or planning to become pregnant during the course of the trial, and patients with other conditions associated with fluctuation of hormones that could lead to refractive changes.

4.3.24 Patients who actively participate in contact sports (i.e., boxing, martial arts) where impacts to the face and eye are a normal occurrence.

4.3.25 Patients participating in any other ophthalmic or non-ophthalmic drug/device clinical trials during the time of this clinical investigation.

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Uncorrected Visual Acuity | 24 months
  After the inlay procedure, patients will attain functional near visual acuity in the inlay eye and functional distance acuity binocularly.

SECONDARY OUTCOMES:
Incidence of Corneal Reaction | 24 months
  Patients treated with low dose mitomycin C will have minimal levels of corneal reaction.
Endothelial Cell Count (measured by Konan Specular Microscope) | 24 months
  Patients treated with low dose mitomycin C will not lose more than 10% of their endothelial cell count from the preoperative measurement

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Whitman, M.D., Principal Investigator — Key-Whitman Eye Center
Locations (3):
- United States (3):
  - Chu Vision Institue, Bloomington, Minnesota
  - Key-Whitman Eye Center, Dallas, Texas
  - Parkhurst NuVision, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No